CLINICAL TRIAL: NCT00949715
Title: Optimize RV Follow-up Selective Site Pacing Clinical Trial
Acronym: ORVFUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Optimize RV Follow-Up
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Results first posted 2013-10-01 (Estimated); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Pacing; Right Ventricular Pacing; Left Ventricular Ejection Fraction
Keywords: Pacemaker; Implantable Pulse Generator (IPG); AV Conduction Disturbance; Selective Site Pacing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RV Mid-Septal Pacing (Active Comparator): Pacing lead located in the right ventricle at the middle of the muscle separating the right and left sides of the heart
  Interventions: Device: Medtronic or Vitatron Dual-Chamber Pacemaker; Device: Medtronic SelectSecure 3830 Lead
- RV Apical Pacing (Active Comparator): Pacing lead located at the bottom of the right ventricle of the heart, in the right ventricular apex
  Interventions: Device: Medtronic or Vitatron Dual-Chamber Pacemaker; Device: Medtronic SelectSecure 3830 Lead

INTERVENTIONS:
Device: Medtronic or Vitatron Dual-Chamber Pacemaker — A Medtronic or Vitatron market-approved dual-chamber implantable pulse generator (IPG) with atrial tachycardia/atrial fibrillation (AT/AF) trending ability
Device: Medtronic SelectSecure 3830 Lead — Medtronic market-approved SelectSecure Model 3830 bipolar pacing lead

SUMMARY:
The purpose of the Optimize RV Follow-Up study is to determine the long-term effect of selective site pacing. Selective site pacing refers to which area of the right ventricle the lead is placed. The goal of selective site pacing is to improve how the heart contracts when paced.

DETAILED DESCRIPTION:
The Optimize RV Follow-Up Selective Site Pacing Clinical Trial is open to subjects that were previously enrolled in the Optimize RV Selective Site Pacing Clinical Trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects enrolled in the Optimize RV study (version 3, dated 6 March 2007)
* Subjects or legal guardians who are willing and able to sign an Informed Consent (and Authorization to use and Disclose Health Information Form, if applicable)

Exclusion Criteria:

* Subjects who have a device that was programmed outside the Optimize RV programming requirements
* Subjects implanted with and implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy (CRT) device
* Subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Optimize RV Follow-Up Team, Study Chair — Medtronic
Locations (12):
- United States (10):
  - Des Moines, Iowa
  - Silver Spring, Maryland
  - Southfield, Michigan
  - Saint Paul, Minnesota
  - New York, New York
  - Cleveland, Ohio
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Tomball, Texas
  - Burlington, Vermont
- Ramat Gan, Israel
- Rovigo, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was open to subjects that were previously enrolled in the original randomized Optimize RV Selective Site Pacing Clnical Trial (ORV)(NCT00422669) who consented between October 2009 through April 2011
Pre-assignment Details: Two of 67 subjects were excluded due to non-compliant programming.
Groups:
- RV Apical Pacing: Pacing lead located at the bottom of the right ventricle of the heart, in the right ventricular apex
  Medtronic or Vitatron Dual-Chamber Pacemaker : A Medtronic or Vitatron market-approved dual-chamber implantable pulse generator (IPG) with atrial tachycardia/atrial fibrillation (AT/AF) trending ability
  Medtronic SelectSecure 3830 Lead : Medtronic market-approved SelectSecure Model 3830 bipolar pacing lead
- RV Mid-Septal Pacing: Pacing lead located in the right ventricle at the middle of the muscle separating the right and left sides of the heart
  Medtronic or Vitatron Dual-Chamber Pacemaker : A Medtronic or Vitatron market-approved dual-chamber implantable pulse generator (IPG) with atrial tachycardia/atrial fibrillation (AT/AF) trending ability
  Medtronic SelectSecure 3830 Lead : Medtronic market-approved SelectSecure Model 3830 bipolar pacing lead
Period: Overall Study
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing
Started | 32 | 33
Completed | 28 | 33
Not Completed | 4 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Missing 24 month LVEF measurement | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.6 (7.6) | 73.3 (10.6) | 74.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 7 | 13 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mean Left Ventricular Ejection Fraction (LVEF) Between RV Pacing Sites at 24 Month
Description: Difference in mean LVEF between pacing sites (RV mid-septal minus RV apex) at 24 months using the 4 chamber view
Time Frame: 24 months
Population: Subjects who had LVEF measurements from both baseline and 24 month timepoints
Measure: Mean (95% Confidence Interval); unit: percentage of LVEF
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing
Number analyzed (Participants) | 28 | 33
percentage of LVEF | 48.3 [43.7 to 53.0] | 51.2 [46.5 to 56.0]
Statistical Analysis 1: Comparison: RV Apical Pacing vs RV Mid-Septal Pacing; HO: Pacing at selective RV sites (mid-septum or apex) has no different impact on the change in LVEF after 24 months follow-up. With 12% SD and 80 subjects in groups will have 90% power to detect an absolute difference in LVEF of 6.2% at 24 months follow-up at an alpha level of 0.05; Test type: Superiority or Other; p = 0.2352, t-test, 2 sided; Mean Difference (Final Values) = 4.0, 95% CI 2-sided [-2.7 to 10.8]

2. Secondary Outcome: Compare the Change in LVEF From the 2 Week Visit (Collected in Prior Study) to the 24 Month Follow-up Visit Between the Optimize RV Mid-Septum Pacing (RVS) Group and RV Apical Pacing (RVA) Group.
Description: Compare the change in LVEF (in the 4 chamber view) from 2 weeks to 24 months between the Optimize RV Mid-Septum Pacing (RVS) group and RV Apical Pacing (RVA) group.
Time Frame: 24 months
Population: Patients that had both 2 week and 24 month follow-up echo data with a 4 chamber LVEF measurement
Measure: Mean (95% Confidence Interval); unit: percentage of LVEF
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing
Number analyzed (Participants) | 28 | 29
percentage of LVEF | -13.5 [-17.7 to -9.2] | -14.6 [-19.7 to -9.4]
Statistical Analysis 1: Comparison: RV Apical Pacing vs RV Mid-Septal Pacing; Ho: Packing at selective RV sites (mid-Septum or apex) has no different impact on LVEF change from 2 weeks to 24 months; Test type: Superiority or Other; p = 0.7405, t-test, 2 sided; Mean Difference (Net) = -1.1, 95% CI 2-sided [-7.6 to 5.5]

3. Secondary Outcome: Compare Change in LV End Systolic Volume After 24 Months Follow-up Between the Optimize RVS Group and RVA Group.
Description: Compare change in 4 chamber LV end systolic volume between baseline and 24 month visit between the Optimize RVS group and RVA group.
Time Frame: 24 months
Population: All subjects who had 4 chamber LV end systolic volume at both the baseline and the 24 month time points
Measure: Mean (95% Confidence Interval); unit: mL
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing
Number analyzed (Participants) | 28 | 33
mL | 55.0 [43.7 to 66.4] | 43.7 [35.0 to 52.4]
Statistical Analysis 1: Comparison: RV Apical Pacing vs RV Mid-Septal Pacing; Ho: Pacing at selective sites (RVS or RVA) has no different impact on LV end systolic volume; Test type: Superiority or Other; p = 0.1051, t-test, 2 sided; Mean Difference (Net) = -11.3, 95% CI 2-sided [-25.1 to 2.4]

4. Secondary Outcome: Compare AT/AF Burden From Baseline to 24 Months Follow-up Between the Optimize RV Mid-Septal (RVS) and RV Apex (RVA) Groups.
Description: Test the difference in AT/AF burden (defined as total duration of minutes in AT or AF relative to total patient follow-up days from baseline to 24 months follow-up) between the Optimize RVS and RVA groups. The proportion can be interpreted as the average time per day that patieents were in AT/AF as collected in the time period from baseline to 24 month follow-up.
Time Frame: Whole time from baseline to 24 months averaged by day
Population: All subjects who meet inclusion/exclusion criteria for the study.
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | RV Apical Pacing | RV Mid-Septal Pacing
Number analyzed (Participants) | 32 | 33
minutes per day | 59.2 (235.3) | 49.3 (199.5)
Statistical Analysis 1: Comparison: RV Apical Pacing vs RV Mid-Septal Pacing; Ho: The AT/AF burden in the RVS group is the same as the RVA group; Test type: Superiority or Other; p = 0.9835, Wilcoxon (Mann-Whitney) — Adjusting for age and gender; Rank Sum; Mean Difference (Net) = 9.9

ADVERSE EVENTS:
Description: The collection of adverse events and subject deaths was not required to meet the objectives of this study and thus was not performed. The products are market approved and used within labeling. Any alleged device related deaths, serious injury, compliants, event would be reported not to this study but via Medical Device Reporting.
Groups:
- No Subjects: No subjects had adverse events or death collected as part of this study.
Arm/Group | No Subjects
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Since the enrollment goal of the study (n=160) was not met (it was decided to stop enrollments after 67 due to slow enrollments), the results of the study were not powered and the results for the primary objective are inconclusive at this time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less